CLINICAL TRIAL: NCT04619797
Title: A Phase II/III, Randomized, Double-Blind, Placebo-Controlled Study of Tiragolumab in Combination With Atezolizumab Plus Pemetrexed and Carboplatin/Cisplatin Versus Pembrolizumab Plus Pemetrexed and Carboplatin/Cisplatin in Patients With Previously Untreated Advanced Non-Squamous Non-Small-Cell Lung Cancer
Brief Title: A Study of Tiragolumab in Combination With Atezolizumab Plus Pemetrexed and Carboplatin/Cisplatin Versus Pembrolizumab Plus Pemetrexed and Carboplatin/Cisplatin in Participants With Previously Untreated Advanced Non-Squamous Non-Small Cell Lung Cancer
Acronym: SKYSCRAPER-06
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO42592; 2020-002851-39 (EudraCT Number); 2022-502031-20-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-30; First posted 2020-11-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Tiragolumab; atezolizumab; Pemetrexed; Carboplatin; Cisplatin; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tiragolumab+Atezolizumab+Pemetrexed+Carboplatin or Cisplatin (Experimental): Induction treatment with tiragolumab in combination with atezolizumab plus pemetrexed and cisplatin or carboplatin will be administered to participants on Day 1 of each 21-day cycle for 4 cycles. Following the induction phase, participants will continue maintenance therapy with tiragolumab in combination with atezolizumab and pemetrexed on Day 1 of each 21-day cycle.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin
- Placebo+Pembrolizumab+Pemetrexed+Carboplatin or Cisplatin (Placebo Comparator): Induction treatment with placebo in combination with pembrolizumab plus pemetrexed and cisplatin or carboplatin will be administered to participants on Day 1 of each 21-day cycle for 4 cycles. Following the induction phase, participants will continue maintenance therapy with placebo in combination with pembrolizumab and pemetrexed on Day 1 of each 21-day cycle.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Tiragolumab Matching Placebo; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab at a fixed dose of 600 milligrams (mg), administered by intravenous (IV) infusion, every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Other Names: MTIG7192A
  Arms: Tiragolumab+Atezolizumab+Pemetrexed+Carboplatin or Cisplatin
Drug: Atezolizumab — Atezolizumab at a fixed dose of 1200 mg, administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Tiragolumab+Atezolizumab+Pemetrexed+Carboplatin or Cisplatin
Drug: Pemetrexed — Pemetrexed 500 milligrams per square meter (mg/m^2), administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
Drug: Carboplatin — Carboplatin at dose of area under the concentration-time curve (AUC) of 5, administered by IV infusion, Q3W on Day 1 of each 21-day cycle for 4 cycles.
Drug: Cisplatin — Cisplatin 75 mg/m^2, administered by IV infusion, Q3W on Day 1 of each 21-day cycle for 4 cycles.
Drug: Tiragolumab Matching Placebo — Matching placebo, administered by IV infusion, Q3W on Day 1 of each 21-day cycle.
  Arms: Placebo+Pembrolizumab+Pemetrexed+Carboplatin or Cisplatin
Drug: Pembrolizumab — Pembrolizumab at a fixed dose of 200 mg, administered by IV infusion, Q3W, on Day 1 of each 21-day cycle.
  Arms: Placebo+Pembrolizumab+Pemetrexed+Carboplatin or Cisplatin

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of tiragolumab in combination with atezolizumab plus pemetrexed and carboplatin/cisplatin (Arm A) compared with placebo in combination with pembrolizumab plus pemetrexed and carboplatin/cisplatin (Arm B) in participants with previously untreated, locally advanced unresectable or metastatic non-squamous non-small cell lung cancer (NSCLC).

Eligible participants will be randomized in a 1:1 ratio to receive one of the following treatment regimens during the induction phase:

* Arm A: Tiragolumab plus atezolizumab plus pemetrexed and carboplatin or cisplatin
* Arm B: Placebo plus pembrolizumab plus pemetrexed and carboplatin or cisplatin

Following the induction phase, participants will continue maintenance therapy with either tiragolumab in combination with atezolizumab and pemetrexed (Arm A) or placebo in combination with pembrolizumab and pemetrexed (Arm B).

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Histologically or cytologically documented locally advanced unresectable or metastatic non-squamous NSCLC that is not eligible for curative surgery and/or definitive chemoradiotherapy
* No prior systemic treatment for metastatic non-squamous NSCLC
* Known tumor programmed death-ligand 1 (PD-L1) status
* Measurable disease, as defined by Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1)
* Life expectancy >= 12 weeks
* Adequate hematologic and end-organ function
* Negative human immunodeficiency virus (HIV) test at screening
* Serology test negative for active hepatitis B virus or active hepatitis C virus at screening.

Key Exclusion Criteria:

* Mutations in epidermal growth factor receptor (EGFR) gene or anaplastic lymphoma kinase (ALK) fusion oncogene
* Pulmonary lymphoepithelioma-like carcinoma subtype of NSCLC
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis
* History of malignancy other than NSCLC within 5 years prior to randomization, with the exception of malignancies with a negligible risk of metastasis or death
* Severe infection within 4 weeks prior to initiation of study treatment or any active infection that, in the opinion of the investigator, could impact patient safety
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T lymphocyte-associated protein 4, anti-TIGIT, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment
* Known allergy or hypersensitivity or other contraindication to any component of the chemotherapy regimen the participant may receive during the study
* Women who are pregnant, or breastfeeding
* Known targetable c-ROS oncogene 1 (ROS1) or BRAFV600E genomic aberration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
Investigator-Assessed Confirmed Objective Response Rate (ORR) (Phase 2) | Up to approximately 5 years
Investigator-Assessed Progression-Free Survival (PFS) (Phase 2 and Phase 3) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
Overall Survival (Phase 3) | From randomization to death from any cause (up to approximately 5 years)

SECONDARY OUTCOMES:
Overall Survival (Phase 2) | From randomization to death from any cause (up to approximately 5 years)
PFS as Determined by an Independent Review Facility (IRF) (Phase 3) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
Investigator-assessed PFS in Participants With PD-L1 Expression at TC ≥50% and TC ≥1% Cut-off, as Determined by Central Testing With Ventana PD-L1 (SP263) Assay (Phase 3) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
OS in Participants With PD-L1 Expression at TC ≥50% and TC ≥1% Cut-off, as Determined by Central Testing With Ventana PD-L1 (SP263) Assay (Phase 3) | From randomization to death from any cause (up to approximately 5 years)
Investigator-Assessed PFS at 6 Months and 12 Months (Phase 3) | 6 months, 12 months
OS Rate at 12 Months and 24 Months (Phase 3) | 12 months, 24 months
Investigator-Assessed Confirmed ORR (Phase 3) | Up to approximately 5 years
Investigator-Assessed Duration of Response (DOR) (Phase 2 and Phase 3) | From first occurrence of a documented confirmed objective response to the first occurrence of disease progression or death from any cause, whichever occurs first (up to approximately 5 years)
Time to Confirmed Deterioration (TTCD) in Participant-Reported Physical Functioning and Global Health Status (GHS)/Quality of Life (QoL) as Measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 (Phase 2 and Phase 3) | Up to approximately 5 years
  TTCD using EORTC Quality-of-Life Questionnaire Core 30 (QLQ-C30) is an initial 10-point decrease in GHS and physical functioning from baseline that must be held for at least two consecutive assessments or an initial clinically meaningful decrease above baseline followed by death. EORTC QLQ-C30: a self-reported measure, consisting of 30 questions that assess 5 aspects of participants functioning (physical, emotional, role, cognitive and social), 3 symptom scales (fatigue, nausea/vomiting and pain), GHS and QoL, and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) with a recall period of the previous week. Functioning items are scored on a 4-point scale: 1=Not at all to 4=Very much, with higher score indicating worse outcome. Symptom items (GHS and QoL) are scored on a 7-point scale: 1=Very poor to 7=Excellent. Scores will be linearly transformed with a minimum score of 0 and maximum score of 100. Higher score indicates better outcome.
TTCD in Participant-Reported Lung Cancer Symptoms for Cough, Dyspnea, and Chest Pain, as Measured by EORTC QLQ-LC13 (Phase 2 and Phase 3) | Up to approximately 5 years
  TTCD using EORTC Quality-of-Life Questionnaire Lung Cancer Module (QLQ-LC13) is an initial 10-point increase in symptom score from baseline that must be held for at least two consecutive assessments or an initial clinically meaningful decrease above baseline followed by death. EORTC QLQ-LC13 consists of 13 lung cancer specific items and includes 11 disease-specific scales/items (dyspnea, coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, pain in chest, pain in arm or shoulder, pain in other parts, pain medication). Each item is scored on a 4-point scale of 1=Not at all to 4=Very much. Scores will be linearly transformed to a score range of 0 to 100. Higher score indicates worsening of symptoms.
Percentage of Participants With Adverse Events (AEs) (Phase 2 and Phase 3) | Up to approximately 5 years
Participants' Response to Side Effects of Treatment as Assessed by EORTC IL46 (Phase 2 and Phase 3) | Up to approximately 5 years
  EORTC Item List 46 (IL46) is a validated single-item question that assesses overall side effect impact. Each item is scored on a 4-point scale of 1=Not at all to 4=Very much. Scores will be linearly transformed to a score range of 0 to 100. Higher score indicates a worse outcome.
Serum Concentration of Tiragolumab (Phase 2 and Phase 3) | Cycle 1 (each cycle=21 days), Day 1: predose, 0.5 hour (h) postdose; Cycles 2, 3, 4, 8, 12, 16, Day 1: predose and at treatment discontinuation (TD) visit (up to approximately 5 years)
Serum Concentration of Atezolizumab (Phase 2 and Phase 3) | Cycle 1 (each cycle=21 days), Day 1: predose, 0.5 hour (h) postdose; Cycles 2, 3, 4, 8, 12, 16, Day 1: predose and at TD visit (up to approximately 5 years)
Percentage of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab (Phase 2 and Phase 3) | Predose on Day 1 of Cycles (each cycle=21 days) 1, 2, 3, 4, 8, 12, 16 and at TD visit (up to approximately 5 years)
Percentage of Participants With ADAs to Atezolizumab (Phase 2 and Phase 3) | Predose on Day 1 of Cycles (each cycle=21 days) 1, 2, 3, 4, 8, 12, 16 and at TD visit (up to approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (128):
- United States (11):
  - UCLA, Los Angeles, California
  - PIH Health Whittier Hospital, Whittier, California
  - SCRI Florida Cancer Specialists South, Fort Myers, Florida
  - SCRI Florida Cancer Specialists North, St. Petersburg, Florida
  - Advent Health Orlando, Winter Park, Florida
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Belgium (4):
  - AZORG Campus Aalst-Moorselbaan, Aalst
  - Cliniques Universitaires St-Luc, Brussels
  - CHU UCL Mont-Godinne, Mont-godinne
  - Vitaz, Sint-Niklaas
- Brazil (7):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - Oncocentro Belo Horizonte, Belo Horizonte, Minas Gerais
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
- China (15):
  - Beijing Cancer Hospital, Beijing
  - Jilin Cancer Hospital, Changchun
  - Xiangya Hospital Central South University, Changsha
  - Affiliated Hospital of Chengde Medical University, Chengde
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital - Sichuan University, Chengdu
  - Anhui Provincial Hospital, Hefei
  - Jinan Central Hospital, Jinan
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Central Hospital, Qingdao
  - Weifang People's Hospital, Weifang
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Denmark (3):
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Onkologisk Afdeling R, Odense C
  - Sjællands Universitetshospital, Roskilde, Roskilde
- France (5):
  - Institut Bergonie, Bordeaux
  - Hopital Nord, Marseille
  - Hopital de Pontchaillou, Rennes
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Larrey, Toulouse
- Germany (5):
  - Helios Klinikum Emil von Behring GmbH, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - St. Vincentius Kliniken Karlsruhe, Karlsruhe
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Medizinische Klinik, Pneumologie, Mainz
  - Klinikum der Philipps-Universität Marburg, Marburg
- Hong Kong (4):
  - Hong Kong United Oncology Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin
- Italy (3):
  - Centro Di Riferimento Oncologico, Aviano, Friuli Venezia Giulia
  - A.O. Villa Scassi, Genoa, Liguria
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
- Japan (13):
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Takarazuka City Hospital, Hyōgo
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Sendai Kousei Hospital, Miyagi
  - Osaka International Cancer Institute, Osaka
  - Kansai Medical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - NHO Kinki Chuo Chest Medical Center, Osaka
  - Saitama Cancer Center, Saitama
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Wakayama Medical University Hospital, Wakayama
- Mexico (4):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Cuidados oncologicos, Querétaro City, Querétaro
  - Oncologico Potosino, San Luis Potosí City, San Luis Potosí
  - ARKE Estudios Clínicos S.A. de C.V., Mexico City
- New Zealand (3):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Waikato Hospital - Cancer and Blood Research Trials Unit, Hamilton
  - Palmerston North Hospital, Palmerston North
- Poland (2):
  - Centrum Terapii Wspolczesnej J.M.Jasnorzewska Spolka Komandytowo-Akcyjna, Lódz
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
- South Korea (10):
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - St. Vincent's Hospital, Gyeonggi-do
  - Samsung Changwon Hospital, Gyeongsangnam-do
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Spain (11):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - ICO L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario Insular?Materno Infantil, Las Palmas de Gran Canaria, LAS Palmas
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Lucus Augusti, Lugo
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (3):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Graubünden Medizin Onkologie, Chur
  - UniversitätsSpital Zürich, Zurich
- Taiwan (3):
  - Changhua Christian Hospital, Chang-hua
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - Vajira Hospital, Bangkok
  - Chulalongkorn Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (7):
  - Adana Baskent University Medical Faculty, Adana
  - Ankara Bilkent City Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Dicle University Faculty of Medicine, Diyarbakır
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Medeniyet University Goztepe Training and Research Hospital., Kadiköy
- United Kingdom (6):
  - Castle Hill Hospital, Hull
  - Barts & London School of Med, London
  - Guy'S Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing
Supporting Information: Study Protocol, SAP